CLINICAL TRIAL: NCT07284212
Title: A Prospective Multicenter Cohort Study on Surgical Treatment Strategies for Pediatric Mitral Regurgitation
Status: Completed | Type: Observational
Sponsor: China National Center for Cardiovascular Diseases (Other Government)
Responsible Party: Sponsor
Other Study IDs: 2020-FW-MR
Record Dates: First submitted 2025-09-24; First posted 2025-12-16 (Actual); Last update posted 2025-12-16 (Actual); Status verified 2025-12

CONDITIONS: Mitral Regurgitation (MR); Pediatric Cardiac Surgery
Keywords: Mitral Regurgitation; Pediatric Cardiac Surgery; Mitral Valve Repair; Surgical Outcomes
MeSH Terms: conditions — Mitral Valve Insufficiency

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Conventional Group: Those who have undergone conventional mitral valve repair
  Interventions: Procedure: conventional mitral valve repair
- Standardized Group: Those who have undergone standardized mitral valve repair
  Interventions: Procedure: standardized mitral valve repair

INTERVENTIONS:
Procedure: conventional mitral valve repair — Patients undergoing conventional mitral valve repair, including annuloplasty, leaflet cleft closure, chordal transfer, and chordal resection, et al.
  Groups: Conventional Group
Procedure: standardized mitral valve repair — Patients undergoing the standardized mitral valve repair strategy proposed by Professor Li at Fuwai Hospital in 2016, which involves comprehensive exploration and correction of abnormalities at the subvalvular, leaflet, and annular levels.
  Groups: Standardized Group

SUMMARY:
This prospective, multicenter cohort study aims to evaluate the outcomes of surgical repair for pediatric mitral regurgitation (MR) in China. From March 2020 to December 2024, consecutive patients younger than 14 years who underwent mitral valve repair at eight representative congenital heart disease centers were enrolled. Eligible patients were those with at least moderate MR on preoperative echocardiography and no prior mitral valve surgery. Patients with uncorrectable concomitant cardiac anomalies, moderate or greater mitral stenosis, ischemic MR, severe leaflet dysplasia, connective tissue disorders (e.g., Barlow, Marfan), cardiomyopathies, or single-ventricle physiology were excluded.

The primary endpoint is a composite of all-cause mortality, reoperation for cardiovascular causes, or recurrence of moderate-or-severe MR during follow-up. Secondary endpoints include perioperative outcomes such as postoperative hospital stay, intensive care unit stay, mechanical ventilation time, and hospitalization cost.

This study is designed to provide high-quality prospective evidence on the safety, durability, and predictors of surgical repair for pediatric MR in a contemporary, real-world, multicenter setting. The findings may inform surgical decision-making and postoperative management strategies for this rare but challenging population.

ELIGIBILITY:
Inclusion Criteria:

* Age < 14 years
* No prior mitral valve surgery
* Preoperative echocardiography demonstrating moderate or severe mitral regurgitation

Exclusion Criteria:

* Concomitant cardiac malformations unable to be corrected simultaneously
* Moderate or severe mitral stenosis
* Ischemic mitral regurgitation
* Severe leaflet dysplasia precluding adequate coaptation
* Connective tissue disorders(e.g., Barlow's disease, Marfan syndrome)
* Any type of cardiomyopathy
* Single ventricle physiology or common atrioventricular valve

Max Age: 14 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Study Population: Children younger than 14 years with moderate or greater mitral regurgitation undergoing surgical repair at eight representative congenital heart disease centers in China. Eligible patients must not have undergone prior mitral valve surgery and must meet the predefined inclusion and exclusion criteria. The study aims to prospectively evaluate surgical outcomes, durability, and predictors of repair from March 2020 to December 2024, with follow-up completed through September 2025.
Sampling Method: Non-Probability Sample
Enrollment: 427 (Actual)
Dates: Start 2020-03-18 (Actual); Primary Completion 2025-09-20 (Actual); Study Completion 2025-09-20 (Actual)

PRIMARY OUTCOMES:
Composite Primary Endpoint | From date of index surgery until last follow-up (up to 5 years)
  Time-to-first event of any of the following: (a) all-cause mortality; (b) mitral valve reoperation; or (c) recurrence of ≥ moderate mitral regurgitation on transthoracic echocardiography.

SECONDARY OUTCOMES:
Postoperative Hospital Length of Stay | perioperatively
  Total postoperative days from surgery to hospital discharge.
ICU Length of Stay | perioperatively
  Consecutive time in intensive care unit.
Duration of Invasive Mechanical Ventilation | perioperatively
  Cumulative duration of invasive mechanical ventilation during the index hospitalization, including all episodes of intubation and re-intubation.
Hospitalization Cost | perioperatively
  Total in-hospital medical cost for the index surgical admission (local currency), extracted from billing records.

CONTACTS AND LOCATIONS:
Locations (1):
- Pediatric Cardiac Surgery Center, Fuwai Hospital, Beijing, Beijing Municipality, China

IPD SHARING:
Plan to Share IPD: No
The data underlying this article cannot be shared publicly for the privacy of individuals that participated in the study.